CLINICAL TRIAL: NCT00910702
Title: The Exploratory Clinical Trials for the Feasibility, Primary Safety and Efficacy of Foldable Capsular Vitreous Body
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: GuangZhou WeiShiBo Biotechnology Co., ltd (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISBOR-61165995
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Retinal Detachment
Keywords: retinal detachment, vitreous body substitute
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FCVB team (Experimental): the vitreous cavity is tamponaded with the foldable capsular vitreous body (FCVB)
  Interventions: Device: foldable capsular vitreous body(FCVB)

INTERVENTIONS:
Device: foldable capsular vitreous body(FCVB) — the vitreous cavity is tamponaded with the foldable capsular vitreous body (FCVB) after PPV
  Other Names: FCVB

SUMMARY:
The purpose of this study is to determine the feasibility, primary safety and efficacy of foldable capsular vitreous body (FCVB) in the treatment of retinal detachment.

DETAILED DESCRIPTION:
Pars plana vitrectomy (PPV) has been one of the most important ophthalmic surgeries for treating a number of blinding diseases by removing and replacing the diseased vitreous body. Current clinic vitreous substitute cannot mimic the natural vitreous which is unable to regenerate after surgery. We have devised a novel foldable capsular vitreous body (FCVB) consisting of a vitreous-like capsule with a tube-valve system, and demonstrated it could finely mimic the morphology and restore main physiological function of the natural vitreous body in our previous study.

ELIGIBILITY:
Inclusion Criteria:

1. Refractive error less than ±3D
2. Visual acuity worse than finger count
3. Ocular perforating injuries, traumatic retinal detachment, giant retinal tear with PVR, serious than grade D PVR, ocular axial length is 16 to 25mm
4. Signed the informed consent form

Exclusion Criteria:

1. Serious heart, lung, liver and kidney dysfunction
2. Serious eye inflammation
3. Silicone oil filled eyes
4. The contralateral eye is non-functional
5. Patients with diseases that the researchers consider not suitable participated in this clinical trial

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Complete retinal reattach rate at the three years after implantation of the silicone-filled FCVB | three years after implantation of the FCVB
  FCVBs filled with balanced salt solution (BSS) were removed from all 11 cases, however, the risk of retinal redetachment and blindness rises after earlier FCVB removal. Approved by the Sun Yat-sen University Medical Ethics Committee, the removal of the FCVB will be decided by doctors depending on the conditions of eye. The eyes implanted with the silicone oil-filled FCVB are still under observation.

SECONDARY OUTCOMES:
visual acuity, intraocular pressure, axial length, ocular inflammatory response, the number of corneal endothelial, anterior chamber angle and ciliary body change, morphological changes of the ocular and FCVB. | Before surgery, 3days,1 week, 2 weeks, 4 weeks, 8 weeks, 3 months, 6 months, 9 months, 1 year, 1.5 years, 2 years, 2.5 years and 3 years after surgery, and 3 months after the removal of the FCVB
  FCVBs filled with BSS were removed from all 11 cases, however, the risk of retinal redetachment and blindness rises after earlier FCVB removal. Approved by the Sun Yat-sen University Medical Ethics Committee, the removal of the FCVB will be decided by doctors depending on the conditions of eye. The eyes implanted with the FCVB and silicone oil are still under observation.

CONTACTS AND LOCATIONS:
Overall Officials: Qianying Gao, MD,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Gao Q, Mou S, Ge J, To CH, Hui Y, Liu A, Wang Z, Long C, Tan J. A new strategy to replace the natural vitreous by a novel capsular artificial vitreous body with pressure-control valve. Eye (Lond). 2008 Mar;22(3):461-8. doi: 10.1038/sj.eye.6702875. Epub 2007 May 25. PMID 17525767
- [Result] Gao Q, Chen X, Ge J, Liu Y, Jiang Z, Lin Z, Liu Y. Refractive shifts in four selected artificial vitreous substitutes based on Gullstrand-Emsley and Liou-Brennan schematic eyes. Invest Ophthalmol Vis Sci. 2009 Jul;50(7):3529-34. doi: 10.1167/iovs.08-2802. Epub 2009 Mar 5. PMID 19264881
- [Derived] Lin X, Ge J, Gao Q, Wang Z, Long C, He L, Liu Y, Jiang Z. Evaluation of the flexibility, efficacy, and safety of a foldable capsular vitreous body in the treatment of severe retinal detachment. Invest Ophthalmol Vis Sci. 2011 Jan 21;52(1):374-81. doi: 10.1167/iovs.10-5869. PMID 20811065